CLINICAL TRIAL: NCT03440593
Title: Utilization of Indirect Calorimetry for Calculation of Nutritional Goals and Its Effect in Ventilator-free Days and Muscle Thickness in Septic Mechanically Ventilated Patients
Brief Title: Indirect Calorimetry Usage and Effect in Ventilator-free Days and Muscle Thickness in Septic Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Baylor IRB#017-362
Record Dates: First submitted 2018-01-17; First posted 2018-02-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2019-01

CONDITIONS: Sepsis; Critical Illness; Respiratory Failure; Nutrition Disorders; Calorie Deficiency; Diaphragm Injury; Quadriceps Muscle Atrophy
Keywords: sepsis; nutrition; indirect calorimetry; muscle thickness
MeSH Terms: conditions — Sepsis; Critical Illness; Respiratory Insufficiency; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measured Arm (Experimental): Patients allocated to the measured energy expenditure (group M) will receive the intervention. Caloric delivery will target results of IC measurement.
  Interventions: Other: Caloric delivery will target results of IC measurement.
- Estimated Arm (No Intervention): Patients allocated to the estimated energy expenditure (group E) will receive nutrition with caloric intake calculated based on the Penn State equation.

INTERVENTIONS:
Other: Caloric delivery will target results of IC measurement. — The prescribed calories to be delivered will be set to target the measurement obtained from performing indirect calorimetry (IC). IC measures the gas exchange of oxygen consumption and carbon dioxide production to determine the true metabolic needs for cellular respiration. The expenditure of calories will be measured utilizing the gas module incorporated within the General Electric Carescape R860 ventilators.
  Arms: Measured Arm

SUMMARY:
Patients admitted to the ICU with diagnosis of sepsis and requiring mechanical ventilation for at least 24-hours and receiving enteral or parenteral nutrition will be prospectively randomized to one of two arms. Patients allocated to the estimated energy expenditure group will receive nutrition with caloric intake calculated based on the Penn State equation. Patients randomized to the measured group will receive nutrition with caloric intake calculated based on IC measurement present in the GE ventilator. Patients in the estimated group will have IC performed, but these data will not be used for prescription of nutrition. An equal number of beds within the ICU will be allocated to the measured group and the estimated group. The primary objective is to assess whether the utilization of indirect calorimetry for caloric goal calculation results in improvement in muscular structure, and consequent reduction of mechanical ventilation duration in patients with sepsis in comparison to utilizing the Penn State estimation equation for caloric goal calculation. The secondary objective is to assess whether the utilization of indirect calorimetry for caloric goal calculation results in improved adequacy of nutritional delivery in comparison to the adequacy of nutritional delivered when utilizing the Penn State estimation equation. Adult patients (> 18 years of age) admitted to the hospital with diagnosis of sepsis, and who require mechanical ventilation during hospitalization will be considered. Patients newly ventilated for at least one day but less than three days will be included in the study. Informed consent will be obtained from the legal authorized representative (LAR).

DETAILED DESCRIPTION:
Mechanically ventilated septic patients admitted to the ICU receiving enteral and or parenteral nutrition will be randomly allocated to one of the aforementioned groups. Demographic information, parameters obtained from the ventilator, muscle measurements through ultrasonography, and clinical information, such as time spent on the mechanical ventilation, time spent in ICU and in the hospital will be collected. Participants will enroll in the study upon admission to the ICU until one of the following occurs-patient is extubated, discharged from the ICU, or death with a maximum of 14 days of ICU admission. Upon inclusion, IC will be assessed at baseline in all patients and then twice weekly. Bedside ultrasonography of the diaphragm and quadricep muscle thickness will be performed upon enrollment of the study (within 3 days of MV and within 1 day of study enrollment) and repeated every 3-5 days with a minimum of twice weekly while on the MV. Severity of illness score (APACHE IV), cause of sepsis, ventilator data, such as average tidal volumes and plateau pressures, cumulative and equivalent doses of sedatives (propofol, midazolam, lorazepam) and analgesics (fentanyl, hydromorphone) will be collected. Presence of delirium during ventilation, based on ICU-CAM scores will be included, as well.

ELIGIBILITY:
Inclusion Criteria:

* New Medical ICU admits
* Mechanically ventilated for one day and less than 3 days upon enrollment
* Adults 18 years or older
* Expected length of ICU stay greater than 3 days
* Initiated on nutrition support (parenteral/or enteral nutrition)
* Sepsis diagnosis documented by physician within one day of ICU admit
* Signed informed consent

Exclusion Criteria:

* Does not meet all criteria of valid indirect calorimetry test for baseline -measurement
* Receiving pulmonary inhaled vasodilator
* Extracorporeal Membrane, Oxygenation (ECMO)
* Pregnancy
* Patients required to be in prone position
* Reintubation
* DNR/AND
* Prisoner
* Employee of BSWH
* Students in contractual agreement with BSWH entity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Ventilator free days (VFD) | From current hospital admission date until the date of hospital discharge, date of death from any cause, whichever came first, assessed up to 28 days.
  The number of days from day 1 to day 28 (of hospital admission) on which the patient was not on the mechanical ventilator. If the patient expired or requires more than 28 days of mechanical ventilation, the value is zero.

SECONDARY OUTCOMES:
Calorie and protein adequacy | Nutritional adequacy will be assessed from day one of ventilation in all patients until extubation from the MV or date of death, whichever came first, assessed up to 14 days.
  Nutritional adequacy of caloric and protein delivery is measured as a ratio of the calories and protein received by the patient compared to the calories and protein prescribed during mechanical ventilation. The ratios are determined individually for calories and protein.
Change in quadricep muscle thickness | Quadricep muscle thickness will be measured upon enrollment to the study (within 72 hours of MV) and every 3-5 days with a minimum of two times per 7 days until extubation from the MV or date of death, whichever came first, assessed up to 14 days.
  Evaluation of the change in muscle thickness during study enrollment in correlation with the adequacy of nutrition delivery.
Change in diaphragm muscle thickness | Diaphragm muscle thickness will be measured upon enrollment to the study (within 72 hours of MV) and then every 3-5 days with a minimum of two times per 7 days until extubation from the MV or date of death, whichever came first, assessed up to 14 days.
  Evaluation of the change in muscle thickness during study enrollment in correlation with the adequacy of nutrition delivery.

OTHER OUTCOMES:
Hospital Mortality | From current hospital admission date until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 24 months.
  Expiration of the participant will be classified as "yes" if patient expired during the current hospital admission.
Hospital length of stay | From current hospital admission date until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 24 months.
  Total number of days patient was admitted to the hospital for the current admission.
Intensive care unit length of stay | From current hospital admission date until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 24 months.
  Total number of days patient was admitted in the intensive care unit for the current hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Mullins, MS, Study Chair — Baylor Health Care System; Ariel Modrykamien, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No